CLINICAL TRIAL: NCT02874079
Title: Genetic Susceptibility and Influence of the Microbiomae in Bullous Pemphigoid
Acronym: MICROPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO15125
Record Dates: First submitted 2016-08-11; First posted 2016-08-22 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Blood Specimen Collection

ARMS (2):
- bullous pemphigoid (Experimental): patients with bullous pemphigoid
  Interventions: Other: Blood sample and cotton skin swabs
- no bullous pemphigoid (Active Comparator): patients with basal cell carcinoma or squamous cell carcinoma and without inflammatory skin disease
  Interventions: Other: Blood sample and cotton skin swabs

INTERVENTIONS:
Other: Blood sample and cotton skin swabs

SUMMARY:
Autoimmune bullous dermatoses include pemphigus, bullous pemphigoid, pemphigoid gestationis, linear IgA dermatosis, mucous membrane pemphigoid, lichen planus pemphigoid, anti-p200 pemphigoid, epidermolysis bullosa acquisita and dermatitis herpetiformis. Autoimmune bullous dermatoses are rare and have an incidence of 20-60 new cases per 1 million person- year in Europe. The incidence of the individual entities is slight significantly different within Europe, but strongly also in comparison to other countries such as Kuwait, Singapore, USA and South America. The most common of these disorders is the bullous pemphigoid.

A considerable progress has been made in the last years to elucidate the pathogenic role of autoantibodies in these diseases. To this end, various in vitro and animal experiments have been used to understand some basic pathophysiological mechanisms in these diseases. Further studies are currently being carried out to explain a precise elucidation of the disease process and to be able to treat the patients targeted later.

At present, however, no data are available to explain why certain individuals develop the autoimmune disease and others do not. Epidemiological studies showed some triggers to the development of autoimmune dysregulation, e.g. drugs.

Furthermore, it has been shown that genetic factors play a role in the pathogenesis of the disease. A clear association with certain HLA regions have been shown in patients with pemphigus, e.g. about 95% of pemphigus patients from the group of Ashkenazi Jews have the HLA-DRB1*0402 haplotype. Recently, the first non-HLA gene associated with pemphigus was described. For other conditions such as bullous pemphigoid, pemphigoid gestationis or linear IgA dermatosis the association with HLA antigens is less pronounced. Another indication of the importance of the genetic background in these diseases can be elucidated from the observation of autoantibodies at a low concentration in healthy relatives of pemphigus patients.

DETAILED DESCRIPTION:
Study genetic and microbiologic predisposition of patients developing a bullous pemphigoid from peripheral blood and skin flora.

ELIGIBILITY:
Inclusion Criteria:

* patients with bullous pemphigoid in active phase
* patients with basal cell carcinoma or squamous cell carcinoma and without inflammatory skin disease
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

- patients with pemphigoid gestationis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
HLA haplotype | Day 1
  the genetic susceptibility in patients bullous pemphigoid were studied by the search of an association between bullous pemphigoid and a particular HLA haplotype

SECONDARY OUTCOMES:
micro satellite markers | Day 1
  the genetic susceptibility in patients bullous pemphigoid were studied by the search of an association between bullous pemphigoid and micro satellite markers, or SNPs (single nucleotide polymorphisms)
SNPs (single nucleotide polymorphisms) | Day 1
  the genetic susceptibility in patients bullous pemphigoid were studied by the search of an association between bullous pemphigoid and SNPs (single nucleotide polymorphisms)
Skin's Bacteria | Day 1
  Analysis of skin microbiome (type and number of bacteria) of patients with bullous pemphigoid, compared with patients without bullous pemphigoid

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France